CLINICAL TRIAL: NCT00445744
Title: Cyclophosphamide Followed by Intravenous Busulfan as Conditioning for Hematopoietic Cell Transplantation in Patients With Myelofibrosis, Acute Myeloid Leukemia, or Myelodysplastic Syndrome.
Brief Title: Cyclophosphamide and Busulfan Followed by Donor Stem Cell Transplant in Treating Patients With Myelofibrosis, Acute Myeloid Leukemia, or Myelodysplastic Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Joachim Deeg, Investigator, Fred Hutchinson Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2130.00; NCI-2010-00270 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); P01HL036444 (NIH)
Record Dates: First submitted 2007-03-07; First posted 2007-03-09 (Estimated); Results first posted 2018-01-02 (Actual); Last update posted 2018-01-02 (Actual); Status verified 2017-12

CONDITIONS: Adult Acute Myeloid Leukemia in Remission; Adult Acute Myeloid Leukemia With 11q23 (MLL) Abnormalities; Adult Acute Myeloid Leukemia With Del(5q); Adult Acute Myeloid Leukemia With Inv(16)(p13;q22); Adult Acute Myeloid Leukemia With t(15;17)(q22;q12); Adult Acute Myeloid Leukemia With t(16;16)(p13;q22); Adult Acute Myeloid Leukemia With t(8;21)(q22;q22); Childhood Acute Myeloid Leukemia in Remission; Childhood Myelodysplastic Syndromes; de Novo Myelodysplastic Syndromes; Essential Thrombocythemia; Myelodysplastic Syndrome With Isolated Del(5q); Polycythemia Vera; Previously Treated Myelodysplastic Syndromes; Primary Myelofibrosis; Recurrent Adult Acute Myeloid Leukemia; Recurrent Childhood Acute Myeloid Leukemia; Secondary Acute Myeloid Leukemia; Secondary Myelodysplastic Syndromes; Secondary Myelofibrosis; Untreated Adult Acute Myeloid Leukemia; Untreated Childhood Acute Myeloid Leukemia and Other Myeloid Malignancies
MeSH Terms: conditions — Congenital Abnormalities; Thrombocythemia, Essential; Chromosome 5q Deletion Syndrome; Polycythemia Vera; Primary Myelofibrosis; Leukemia, Myeloid, Acute | interventions — Cyclophosphamide; Busulfan; Tacrolimus; Methotrexate; merphos; Cytogenetic Analysis; Flow Cytometry; Pharmacogenomic Testing; Peripheral Blood Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (cyclophosphamide, busulfan, transplant) (Experimental): CONDITIONING REGIMEN: Patients receive cyclophosphamide IV on days -7 and -6 and busulfan IV over 3 hours on days -5 to -2.
  TRANSPLANTATION: Patients undergo allogeneic peripheral blood stem cell transplant on day 0.
  POST-TRANSPLANT IMMUNOSUPPRESSION: Patients receive tacrolimus IV or PO twice daily on days -1 to 200 with taper on day 56 and methotrexate on days 1, 3, 6, and 11.
  Interventions: Drug: cyclophosphamide; Drug: busulfan; Drug: tacrolimus; Drug: methotrexate; Genetic: cytogenetic analysis; Other: flow cytometry; Other: pharmacological study; Other: pharmacogenomic studies; Procedure: peripheral blood stem cell transplantation; Procedure: allogeneic hematopoietic stem cell transplantation

INTERVENTIONS:
Drug: cyclophosphamide — Given IV
  Other Names: CPM; CTX; Cytoxan; Endoxan; Endoxana
Drug: busulfan — Given IV
  Other Names: BSF; BU; Misulfan; Mitosan; Myeloleukon
Drug: tacrolimus — Given IV or PO
  Other Names: FK 506; Prograf
Drug: methotrexate — Given IV
  Other Names: amethopterin; Folex; methylaminopterin; Mexate; MTX
Genetic: cytogenetic analysis — Correlative studies
Other: flow cytometry — Correlative studies
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies
Other: pharmacogenomic studies — Correlative studies
  Other Names: Pharmacogenomic Study
Procedure: peripheral blood stem cell transplantation — Undergo PBPC transplantation
  Other Names: PBPC transplantation; PBSC transplantation; peripheral blood progenitor cell transplantation; transplantation, peripheral blood stem cell
Procedure: allogeneic hematopoietic stem cell transplantation — Undergo allogeneic transplantation

SUMMARY:
This trial is studying the side effects and how well giving cyclophosphamide and busulfan followed by donor stem cell transplant works in treating patients with myelofibrosis, acute myeloid leukemia, or myelodysplastic syndrome. Giving chemotherapy, such as cyclophosphamide and busulfan, before a donor stem cell transplant helps stops the growth of cancer cells. It also helps stop the patient's immune system from rejecting the donor's stem cells. The donated stem cells may replace the patient's immune cells and help destroy any remaining cancer cells (graft-versus-tumor effect). Sometimes the transplanted cells from a donor can also make an immune response against the body's normal cells. Giving tacrolimus and methotrexate after the transplant may stop this from happening

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the incidence of hepatotoxicity with a conditioning regimen of CY (cyclophosphamide)/tBU (busulfan) in patients receiving hematopoietic cell transplant (HCT).

SECONDARY OBJECTIVES:

I. To determine overall and non-relapse mortality at day +200 after HCT.

II. To determine the peak bilirubin levels through day +20 after HCT.

III. To determine the incidence of pulmonary toxicity in the form of idiopathic pulmonary syndrome (IPS).

IV. To determine the rate of graft failure.

V. To determine the time to engraftment.

VI. To determine the rate of relapse.

VII. To determine the incidence and severity of graft-versus-host disease (GVHD).

VIII. To evaluate the pharmacokinetics/dynamics of BU and CY.

X. To evaluate the pharmacogenomics of response, toxicity and pharmacokinetics of CY/tBU.

OUTLINE:

CONDITIONING REGIMEN: Patients receive cyclophosphamide intravenously (IV) on days -7 and -6 and busulfan IV over 3 hours on days -5 to -2.

TRANSPLANTATION: Patients undergo allogeneic peripheral blood stem cell transplant on day 0.

POST-TRANSPLANT IMMUNOSUPPRESSION: Patients receive tacrolimus IV or orally (PO) twice daily on days -1 to 200 with taper on day 56 and methotrexate on days 1, 3, 6, and 11.

After completion of study treatment, patients are followed periodically.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic myelofibrosis (CIMF)
* Myelofibrosis developing with polycythemia vera or essential thrombocythemia
* Acute myeloid leukemia with or without antecedent hematologic disorder, at any disease stage (complete remission, minimal residual disease, or relapsed leukemia)
* Myelodysplastic syndrome of any World Health Organization (WHO) or French-American-British (FAB) category, at any disease stage
* Less than 61 years of age if transplanted from an unrelated donor, or less than 66 years of age if transplanted from a related donor
* Receiving unmanipulated peripheral blood stem cells from an human leukocyte antigen (HLA)-identical or 1-allele-mismatched related or unrelated donor, or receiving G-CSF-stimulated bone marrow if co-enrolled on Fred Hutchinson Cancer Research Center (FHCRC) protocol 2250
* With a Karnofsky Performance score of > 70% at the time of pre-transplant evaluation
* Able to give informed consent (if >= 18 years of age), or with a legal guardian capable of giving consent (if < 18 years of age)
* DONOR: HLA-identical or 1-allele-mismatched related or unrelated donors (by high resolution typing)
* DONOR: Undergoing peripheral blood stem cell harvest or G-CSF-stimulated bone marrow harvest (bone marrow permitted only as part of FHCRC protocol 2250)
* DONOR: In good general health, with a Karnofsky performance score of > 80%
* DONOR: Able to give informed consent (if >= 18 years of age), or with a legal guardian able to give informed consent (if < 18 years of age and donating for a related transplant)

Exclusion Criteria:

* Without an HLA-identical or 1-allele-mismatched related or unrelated donor
* With human immunodeficiency virus (HIV) positivity or active infectious hepatitis
* Receiving a medication known to strongly inhibit enzymes in the CYP450 pathway, and which, in the judgment of the consenting provider, cannot be safely discontinued for the duration of conditioning
* Whose life expectancy is severely limited by diseases other than the hematologic disorder for which they are undergoing HCT (HCT-comorbidity index [CI] > 3)
* Women who are pregnant or lactating
* With known hypersensitivity to BU or CY
* With hepatic dysfunction as evidenced by total bilirubin or AST > 2x the upper limit of normal, or evidence of synthetic dysfunction or cirrhosis
* With impaired renal function, as evidenced by creatinine clearance < 50% of expected, creatinine > 2x the upper limit of normal, or dialysis dependence
* With impaired pulmonary function, as evidenced by pO2 < 70 mm Hg and diffusing capacity of carbon monoxide (DLCO) < 70% predicted or by pO2 < 80 mm Hg and DLCO < 60%, or receiving continuous supplementary oxygen
* With impaired cardiac function, as evidenced by ejection fraction < 35% or active coronary artery disease
* Unable to give informed consent
* DONOR: Deemed unable to undergo stem cell collection, for any reason
* DONOR: HIV-positive, or hepatitis B or C antigen-positive
* DONOR: Women with a positive pregnancy test
* DONOR: Unable to give informed consent (if >= 18 years of age), or without a legal guardian able to give informed consent (if <18 years of age)

Max Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2006-12; Primary Completion 2011-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Rezvani, Principal Investigator — Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Locations (1):
- Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (Cyclophosphamide, Busulfan, Transplant): CONDITIONING REGIMEN: Patients receive cyclophosphamide IV on days -7 and -6 and busulfan IV over 3 hours on days -5 to -2.
  TRANSPLANTATION: Patients undergo allogeneic peripheral blood stem cell transplant on day 0.
  POST-TRANSPLANT IMMUNOSUPPRESSION: Patients receive tacrolimus IV or PO twice daily on days -1 to 200 with taper on day 56 and methotrexate on days 1, 3, 6, and 11.
  cyclophosphamide: Given IV
  busulfan: Given IV
  tacrolimus: Given IV or PO
  methotrexate: Given IV
  cytogenetic analysis: Correlative studies
  flow cytometry: Correlative studies
  pharmacological study: Correlative studies
  pharmacogenomic studies: Correlative studies
  peripheral blood stem cell transplantation: Undergo PBPC transplantation
  allogeneic hematopoietic stem cell transplantation: Undergo allogeneic transplantation
Period: Overall Study
Arm/Group | Treatment (Cyclophosphamide, Busulfan, Transplant)
Started | 52
Completed | 51
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Cyclophosphamide, Busulfan, Transplant)
Number analyzed (Participants) | 51
Age, Continuous [Median (Full Range); unit: years] | 55 [30 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 30

OUTCOME MEASURES:

1. Primary Outcome: Effectiveness of Cyclophosphamide/Busulfan Regimen in Reducing Regimen-related Liver Toxicity
Description: Number of patients with regimen-related liver toxicity. Diagnoses will be made according to the established criteria initially proposed in 1984 by McDonald et al.
Time Frame: Up to day +20
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Cyclophosphamide, Busulfan, Transplant)
Number analyzed (Participants) | 51
Participants | 8

2. Primary Outcome: Non-relapse Mortality (NRM) (Patients With AML/MDS)
Description: Cumulative incidence rate with death as a competing risk, assessed at day 100.
Time Frame: Up to day 200
Measure: Number; unit: percent
Arm/Group | Treatment (Cyclophosphamide, Busulfan, Transplant)
Number analyzed (Participants) | 31
percent | 17

ADVERSE EVENTS:
Time Frame: Up to 3 years after enrollment
Description: Causes of death were recorded as adverse events. Other adverse events were not recorded in this study.
Arm/Group | Treatment (Cyclophosphamide, Busulfan, Transplant)
All-Cause Mortality (participants affected / at risk) | 19/52
Serious Adverse Events (participants affected / at risk) | 19/52
Other Adverse Events (participants affected / at risk) | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Cyclophosphamide, Busulfan, Transplant) (N=52)
graft-versus-host disease (Immune system disorders) | 2
Recurrent or progressive malignancy (Blood and lymphatic system disorders) | 9
Infection associated with graft-versus-host disease (Infections and infestations) | 4
infection not associated with graft-versus-host disease (Infections and infestations) | 2
Secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
suicide (Psychiatric disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No